CLINICAL TRIAL: NCT05492838
Title: Clinical and Radiographic Evaluation of Socket Shield Technique With or Without Flap Elevation
Brief Title: Socket Shield Technique With or Without Flap Elevation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Ezgi Gürbüz, Assist. Prof., Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02
Record Dates: First submitted 2022-08-03; First posted 2022-08-09 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2023-10

CONDITIONS: Alveolar Bone Resorption
Keywords: Socket Shield Technique; Alveolar Bone Preservation; Immediate Implantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flapless Surgery (Active Comparator)
  Interventions: Procedure: Immediate implantation with the Socket Shield Technique
- Surgery With Flap Elevation (Active Comparator)
  Interventions: Procedure: Immediate implantation with the Socket Shield Technique

INTERVENTIONS:
Procedure: Immediate implantation with the Socket Shield Technique — Immediate implant surgery applied with the Socket Shield Technique

SUMMARY:
It is aimed to compare the bone changes and the amount of marginal bone loss after prosthetic loading around the immediately placed implants using the Socket Shield Technique with or without flap elevation.

DETAILED DESCRIPTION:
Temporary prostheses will be applied to patients in the flap and flapless surgery group 1 week after the surgical procedure, and permanent prostheses will be placed 3 months later. From this date, clinical controls will be made in the 1st, 3rd, 6th months and 1st year.

During these controls, biological complications (peri-implant mucositis, peri-implantitis), implant failure and survival rates, and complications related to the socket shield (socket shield exposure, infection) will be evaluated. Marginal bone loss around the implants and bone resorption in the horizontal and vertical directions will be compared between the two groups with cone beam computed tomography taken at the 1st year follow-up.

The Oral Health-Related Quality of Life Scale will be applied in the session where the temporary prosthesis is applied 1 week after the surgery, in the 1st month clinical control and in the 3rd and 6th month clinical control after the permanent prosthesis application, in order to evaluate the quality of life related to the surgical and prosthetic application of the patients in both groups, and comparisons between groups will be made.

In addition, intraoral photographs will be taken from the patients for aesthetic evaluation before the surgical procedure, at the 1st, 3rd and 6th month clinical control sessions. Pink Aesthetic Score (PES) and White Aesthetic Score (BES) will be evaluated on the photographs, and a comparison will be made between groups in terms of scores.

ELIGIBILITY:
Inclusion Criteria:

* Being systemically healthy (ASA classification I-II)
* Being over 18 years old
* Not smoking
* Having good oral hygiene
* Upper incisors and premolars that cannot be restored and have extraction indications
* Periodontally healthy, non-mobile teeth
* The amount and quality of bone suitable for immediate implant placement

Exclusion Criteria:

* Periodontally unhealthy teeth
* Teeth with vertical root fracture on the buccal surface
* Teeth with a horizontal fracture below the bone level
* Teeth with external and internal resorption affecting the buccal part of the root
* Patients who are pregnant or suspected of pregnancy

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2024-12-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline marginal bone loss at 12 months | Baseline, 12th month
  Measurement of marginal bone loss change between baseline and 12th month by cone beam computed tomography

SECONDARY OUTCOMES:
Change of peri-implant pocket depth between baseline and follow-up periods | Baseline, 1st month, 3rd month, 6th month, 12th month
  Clinical measurement of change in peri-implant pocket depth between follow-up periods using probe
Change of modified plaque index between baseline and follow-up periods | Baseline, 1st month, 3rd month, 6th month, 12th month
  Clinical measurement of change in modified plaque index between follow-up periods using probe
Change of modified bleeding index between baseline and follow-up periods | Baseline, 1st month, 3rd month, 6th month, 12th month
  Clinical measurement of change in modified bleeding index between follow-up periods using probe
Change in the width of keratinized mucosa between follow-up periods | Baseline, 1st month, 3rd month, 6th month, 12th month
  Clinical measurement of change in the keratinized mucosa width between follow-up periods using probe
Change in the mucosal recession between follow-up periods | Baseline, 1st month, 3rd month, 6th month, 12th month
  Clinical measurement of change in the mucosal recession between follow-up periods using probe
Change in the mucosal thickness between follow-up periods | Baseline, 1st month, 3rd month, 6th month, 12th month
  Clinical measurement of change in the mucosal thickness between follow-up periods using spreader
Visual analog scale | Baseline, 1st week, 1st month, 3rd month, 6th month, 12th month
  On a scale of 0-10, with 0 indicating the worst and 10 indicating the best choice
Oral health impact profile questionnaire | Baseline, 1st week, 1st month, 3rd month, 6th month, 12th month
  A questionnaire consisting of 14 items
Pink aesthetic score | Baseline, 1st week, 1st month, 3rd month, 6th month, 12th month
  An index with a minimum score of 0 and a maximum score of 14
White aesthetic score | Baseline, 1st week, 1st month, 3rd month, 6th month, 12th month
  An index with a minimum score of 0 and a maximum score of 10

CONTACTS AND LOCATIONS:
Overall Officials: Ezgi Gürbüz, Principal Investigator — Kutahya Health Sciences University
Locations (1):
- Kutahya Health Sciences University, Kütahya, Turkey (Türkiye)